CLINICAL TRIAL: NCT02289937
Title: Effect of a Lateral Nerve of the Thigh Block on Postoperative Pain After Total Hip Replacement Surgery: a Clinical Randomized Trial
Brief Title: Effect of a Lateral Nerve of the Thigh Block on Postoperative Pain After Total Hip Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Hägi-Pedersen (Other)
Responsible Party: Sponsor-Investigator, Daniel Hägi-Pedersen, Consultant, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001-2013; 2013-004501-12 (EudraCT Number)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Pain, Postoperative; Anesthesia, Conduction; Arthroplasty, Replacement, Hip
Keywords: Postoperative pain; regional anaesthesia; total hip replacement; nervus cutaneous femoral lateralis
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): 8 ml of ropivacaine 7,5 mg/ml will be injected around nervus cutaneous femoral lateralis. Ultrasound-guided.
  Interventions: Drug: Ropivacaine; Device: An ultrasound-guided Nervus cutaneous femoral lateralis blockade will be given postoperatively
- Placebo (Placebo Comparator): 8 ml of isotonic saline will be injected around nervus cutaneous femoral lateralis. Ultrasound-guided
  Interventions: Drug: Placebo; Device: An ultrasound-guided Nervus cutaneous femoral lateralis blockade will be given postoperatively

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Placebo
  Other Names: Saline, NaCl
  Arms: Placebo
Device: An ultrasound-guided Nervus cutaneous femoral lateralis blockade will be given postoperatively

SUMMARY:
The purpose of this study was to evaluate the analgesic efficacy of the nervus cutaneous femoral lateralis (NCFL) blockade on postoperative pain after total hip replacement surgery. The NCFL-block is a pure sensory block. We hypothesized that the NCFL-block would reduced the postoperative pain without delaying mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip replacement

Exclusion Criteria:

* general anaesthesia
* Allergy to local anesthetics of the amide type
* Revision surgery
* Bilateral surgery
* Chronic pain patient
* Women in the fertile age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
VAS-score 4 hours postoperative during movement | 4 hours postoperative
  VAS-score 4 hours postoperative during 30 degrees of flexion of the hip. VAS-score: 0-100 mm; 0: no pain, 100: worst imaginable pain.

SECONDARY OUTCOMES:
VAS-score 0-24 hours postoperative during movement | 0-24 hours postoperatively
  VAS-score 0, 1, 2, 8, 12, and 24 hours postoperative during 30 degrees of flexion of the hip. VAS-score: 0-100 mm; 0: no pain, 100: worst imaginable pain.
VAS-score 0-24 hours postoperative at rest | 0-24 hours postoperatively
  VAS-score 0, 1, 2, 4, 8, 12, and 24 hours postoperative at rest. VAS-score: 0-100 mm; 0: no pain, 100: worst imaginable pain.
Oxynorm consumption | 0-24 hours postoperative
  Oxynorm consumption 24 hours postoperative
time to first oxynorm requirement | 0-24 hours postoperatively
Mobilization | 0-24 hours postoperatively
  time to first mobilization
Mobilization | 0-24 hours postoperatively
  Ability to mobilize judged by the cumulated ambulation (CAS) score: 0-6; 0 no mobilization, 6: fully mobilized
Length of stay | 0-7 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hägi-Pedersen, M.D., Ph.D., Study Chair — Naestved Hospital, Department of Anaesthesiology